CLINICAL TRIAL: NCT01453192
Title: National, Multicenter, Phase III Prospective Trial About Clinical and Immunological Follow-up After Renal Transplantation in HIV-1 Infected Patients With End Stage Chronic Renal Insufficiency
Brief Title: Renal Transplantation and Raltegravir in HIV-Infected Patients
Acronym: ANRS153TREVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-001004-35; ANRS 153 TREVE (Registry Identifier: ANRS)
Record Dates: First submitted 2011-10-03; First posted 2011-10-17 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: HIV-1 Infection; Chronic Renal Insufficiency
Keywords: Raltegravir; Renal transplantation; HIV-1; Acute renal graft rejection
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Raltegravir (Experimental): Raltegravir associated to an antiretroviral regimen without ritonavir boosted antiprotease
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Introduction of Raltegravir 2 days after renal transplantation within an antiretroviral regimen without ritonavir boosted antiprotease
  Other Names: Isentress

SUMMARY:
The aim of this study is to evaluate the incidence of acute renal graft rejection 6 months after transplantation in HIV-infected patients under three antiretroviral drugs regimen including Raltegravir.

DETAILED DESCRIPTION:
Antiretroviral treatment of HIV-1 Infection might interact with immunosuppressive treatments which increase rejection of renal graft incidence.

In addition HIV infection may be modified together with cardiovascular risk. Patients participating to this study will receive after transplantation antiretroviral regimen including Raltegravir.

Raltegravir treatment does not interact with immunosuppressive drugs and thus seems to be the treatment of choice to be associated with immunosuppressive drugs.

ELIGIBILITY:
Inclusion Criteria:

* Registration on the French national renal transplantation waiting list (Biomedicines Agency) for a living or cadaveric donor organ
* HIV-1-infected patients treated by a three-drug ARV regimen
* Immuno-virologic criteria at renal transplantation: undetectable viral load (<50 copies/mL) and CD4 >200/mm3 for at least three months on stable ARV
* Age >18 years and <70 years
* Effective contraception for women
* Written informed consent
* Patient with social security coverage

Exclusion Criteria:

* Permanent:

  * Hepatic cirrhosis
  * Serious psychiatric illness history
  * EBV or HHV8 lymphoproliferation (lymphoma, systemic Kaposi's sarcoma or multifocal Castleman's disease)
  * History of PML
  * HTLV-1 seropositivity
  * Severe pulmonary or cardiovascular disease with poor short-term vital prognosis
  * Patient with AgHBs+
  * History of cryptosporidiosis
  * History of fungal infection with multi resistant fungi not likely to respond to oral antifungal therapy
  * Impossibility or refusal of Raltegravir switch, decision made by doctor or patient
* Temporary:

  * Recent malignancy (between 2 and 5 years according to type)
  * HPV-related cervical or anal disease: carcinoma in situ, AIN III, CIN III in remission for less than three years
  * Active infection
  * HCV infection (PCR-positive)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Incidence of acute clinical renal graft rejection | 6 months
  Incidence of acute clinical renal graft rejection defined by 20% increase of serum creatinine, associated to histological features (Banff classification) 6 months after renal transplantation

SECONDARY OUTCOMES:
Incidence of acute clinical and subclinical renal graft rejection | 1 year
  Incidence of acute clinical and subclinical renal graft rejection up to 1 year after renal transplantation defined only by renal histology (without creatinine modification). Histology is performed on routine renal graft biopsy 3 months and 1 year after transplantation.
One year graft survival | 1 year
  One year graft survival, compared to non HIV-infected transplanted patients, using data provided by French Biomedicines Agency
Patients' survival | 1 year
  Patients survival, compared to:
  - chronic dialysis HIV patients still listed on the transplantation waiting list - transplanted non-HIV patients using data provide by French Biomedicine Agency
Phenotyping of lymphocytic infiltrates in case of acute rejection | 1 year
  The aim of the immunological phenotyping is to analyse the expression of activation markers between different TCD4 and TCD8 sub-population, this phenotyping will be compared to those observed in acute cell-mediated rejection occurring in the historical cohort of Non-HIV patients. In addition, the rate and expression of Treg population will be evaluated.
Incidence of AIDS defined diseases and severe morbidity diseases after renal transplantation | 1 year
  Severe morbidity diseases include: pathological infections, malignancies, metabolic and cardiovascular diseases.
Immunological and virologic status after renal transplantation | 1 year
  Immunological (lymphocyte activation and inflammatory parameters) and virologic status (kinetics of viral replication: HIV RNA in blood, total HIV DNA in PBMC) monitoring after renal transplantation. These parameters will be compared with pre-transplant status.
Evaluation of the switch by raltegravir at the time of renal transplantation | 1 year
  Assessment of ARV medications change and introduction of raltegravir at the time of renal transplantation in terms of reduction of pharmacokinetic interaction between antiretroviral regimen including raltegravir and immunosupressive treatments. In addition, virological efficacy of antiretroviral treatment including Raltegravir will be evaluated.
Viral load control after switch by antiretroviral treatment including raltegravir after renal transplantation | 1 year
  The aim of this study is to evaluate at the time of renal transplantation the virologic efficiency after the switch by an antiretroviral regimen including Raltegravir in terms of viral load control an virological failure as Raltegravir is known for its low genetic barrier.
Survival and waiting period of HIV patients registered on French biomedicine agency for renal transplantation | 1 year
  Assessment of HIV patients' waiting period until renal transplantation and survival of patients registered on French biomedicine agency waiting-list compared to Non-HIV population (data provided by French Biomedicine Agency )
Measurement of Area under plasma concentration (AUC) variability of immunosuppressive drugs after introduction of antiretroviral regimen containing Raltegravir | 1 year
  Area under plasma concentration (AUC) of Raltegravir and immunosuppressive drugs (Tacrolimus and Mycophenolate Mophetyl) will be measured as well as residual concentration of Tacrolimus. This study is performed in order to verify immunosupressive treatments dosage adaptation.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GRIMBERT, MD, Principal Investigator — CHU Henri-Mondor; Dominique COSTAGLIOLA, PHD, Study Director — INSERM U943
Locations (14):
- France (14):
  - Hôpital Pellegrin, Service de Nephrologie, Transplantation Rénale, Dialyse, Bordeaux
  - CHU De Caen, Service de Néphrologie Hémodialyse, Caen
  - Hôpital Henri Mondor, Service de Néphrologie Transplantation, Créteil
  - Hôpital Kremlin Bicêtre, Service de Néphrologie, Le Kremlin-Bicêtre
  - CHRU Lille, Service de néphrologie, Lille
  - CHU de Nantes, Service de Néphrologie et Immunologie Clinique, Nantes
  - Hôpital Pasteur, Service de Néphrologie - Transplantation, Nice
  - Hopital Saint Louis, Service de Néphrologie, Paris
  - Hôpital Necker, Service de Néphrologie adulte, Paris
  - Hôpital TENON, Urgences Néphrologiques et Transplantation Rénale, Paris
  - Hôpital civil, Service de Néphrologie et Transplantation, Strasbourg
  - Hôpital Foch, Service de Néphrologie Transplantation, Suresnes
  - Hôpital Rangueil, Service de Néphrologie, HTA, Dialyse, Transplantation, Toulouse
  - Hôpital Bretonneau, Service de Néphrologie, Tours

REFERENCES:
- See also: French National Agency for Research on AIDS and viral Hepatitis — http://www.anrs.fr